CLINICAL TRIAL: NCT03734705
Title: Efficacy and Feasibility of Intensive Imaginal Exposure for Hoarding Disorder
Brief Title: Imaginal Exposure for Hoarding Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 48109
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hoarding Disorder
Keywords: hoarding disorder; intolerance of uncertainty; experiential avoidance; imaginal exposure; clutter; attachment
MeSH Terms: conditions — Hoarding Disorder; Speech Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomly assigned to imaginal exposure writing intervention or neutral control writing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaginal Exposure Writing (Experimental): People with hoarding disorder will write for 20 minutes on each of 3 consecutive days about their worst-case scenario regarding discarding a possession (i.e., imaginal exposure).
  Interventions: Behavioral: Imaginal Exposure Writing
- Neutral Writing (Sham Comparator): People with hoarding disorder will write for 20 minutes on each of 3 consecutive days about what they would do if they had a day off work or school.
  Interventions: Other: Neutral Writing

INTERVENTIONS:
Behavioral: Imaginal Exposure Writing — Imaginal exposure is a psychotherapy strategy that has been studied and shown to be helpful in the improvement of symptoms (e.g., anxiety, worry) for other psychiatric conditions, including excessive worry and obsessive-compulsive disorder symptoms.
  Arms: Imaginal Exposure Writing
Other: Neutral Writing — Used in prior research as a control condition for imaginal exposure. Neutral writing will involve writing about what one would do on a day off work or school.
  Arms: Neutral Writing

SUMMARY:
The present study will test a potential new treatment strategy, imaginal exposure, for hoarding disorder. Although cognitive behavioral therapy often reduces hoarding, some people do not want to start, or cannot handle, that option. To help such individuals, the present study will provide imaginal exposure therapy to people with hoarding disorder, wherein they imagine discarding possessions as a way of becoming acclimated to the idea. We predict that imaginal exposure will improve hoarding symptoms as well as two psychological experiences linked to the condition: intolerance of uncertainty and emotional avoidance.

DETAILED DESCRIPTION:
Hoarding disorder is a common mental illness characterized by difficulty parting with possessions and by clutter that makes living spaces unusable. Cognitive behavioral therapy (CBT) is an effective treatment for hoarding disorder, but new approaches are needed to engage those who are reluctant to start or cannot tolerate CBT. Both intolerance of uncertainty and emotional avoidance are linked to hoarding disorder and may interfere with treatment engagement. Imaginal exposure, a therapeutic technique which involves repeatedly imagining feared scenarios and experiencing the evoked emotions, effectively targets both intolerance of uncertainty and emotional avoidance. The present study is the first to test whether imagining discarding possessions can improve hoarding symptoms more than does a control exercise. We hypothesize that compared to a control exercise, imaginal exposure will improve hoarding symptoms, intolerance of uncertainty and emotional avoidance.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Any gender and all ethno-racial categories
3. Hoarding Disorder primary condition
4. Willing and able to understand and complete consent and study procedures
5. English speaking

Exclusion Criteria:

1. Severe depression
2. Clinically at risk of suicide with Columbia Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation Subscale of 4 or higher (i.e. suicidal intent without specific plan)
3. Currently receiving Cognitive Behavioral Therapy (CBT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Fracalanza, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fracalanza K, Raila H, Avanesyan T, Rodriguez CI. Written Imaginal Exposure for Hoarding Disorder: A Preliminary Pilot Study. J Nerv Ment Dis. 2024 May 1;212(5):289-294. doi: 10.1097/NMD.0000000000001719. PMID 38598729

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imaginal Exposure Writing | Neutral Writing
Started | 17 | 15
Completed | 17 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imaginal Exposure Writing | Neutral Writing | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.94 (10.74) | 48.33 (15.71) | 52.91 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 10 | 18
  Black | 0 | 0 | 0
  East Asian | 4 | 4 | 8
  Southeast Asian | 0 | 0 | 0
  Latin American | 3 | 0 | 3
  Mixed Race | 2 | 0 | 2
  Other ethnicity | 0 | 1 | 1
Employment Status [Count of Participants; unit: Participants]
  Not working (including student) | 5 | 2 | 7
  Employed (full or part-time) | 9 | 9 | 18
  Retired | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Savings Inventory Revised (Frost, Steketee & Grisham, 2004; Tolin, Meunier, Frost & Steketee, 2011)
Description: Gold-standard 23-item self-report measure of hoarding disorder symptoms. Scale scores range from 0 to 92, with higher scores indicating more severe hoarding symptoms. More severe hoarding symptoms are considered a worse outcome.
Time Frame: Baseline (Pre Writing) and Follow Up (week 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imaginal Exposure Writing | Neutral Writing
Number analyzed (Participants) | 17 | 15
score on a scale
  Pre Writing | 62.41 (13.22) | 62.60 (11.97)
  Follow Up | 53.41 (16.87) | 52.00 (14.05)

2. Secondary Outcome: Compulsive Acquisitions Scale (Frost et al. 2002)
Description: Self-report 18-item measure of behaviors associated with hoarding disorder (i.e., acquiring).Scale scores range from 18 to 126, with higher scores indicating more severe hoarding behaviors. More severe hoarding behaviors are considered a worse outcome.
Time Frame: Baseline (Pre Writing) and Follow Up (week 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imaginal Exposure Writing | Neutral Writing
Number analyzed (Participants) | 17 | 15
score on a scale
  Pre Writing | 62.88 (29.59) | 57.93 (27.68)
  Follow Up | 56.76 (30.47) | 47.47 (23.52)

3. Secondary Outcome: Intolerance of Uncertainty Scale (Buhr & Dugas, 2002)
Description: Self-report 27-item measure of a cognitive process related to hoarding called intolerance of uncertainty. Scale scores range from 27 to 135 (some items are reverse scored), with higher scores indicating more severe intolerance of uncertainty. More severe intolerance of uncertainty is considered a worse outcome.
Time Frame: Baseline (Pre Writing) and Follow Up (week 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imaginal Exposure Writing | Neutral Writing
Number analyzed (Participants) | 17 | 15
score on a scale
  Pre Writing | 68.47 (31.63) | 72.27 (28.86)
  Follow Up | 65.06 (33.27) | 65.47 (30.21)

4. Secondary Outcome: Acceptance and Action Questionnaire - II (Hayes, Luoma, Bond, Masuda and Lillis, 2006)
Description: Self-report 7-item measure of a cognitive process related to hoarding called experiential avoidance. Scale scores range from 7 to 49, with higher scores indicating more severe experiential avoidance. More severe hoarding behaviors are considered a worse outcome.
Time Frame: Baseline (Pre Writing) and Follow Up (week 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imaginal Exposure Writing | Neutral Writing
Number analyzed (Participants) | 17 | 15
score on a scale
  Pre Writing | 24.94 (12.40) | 28.33 (10.93)
  Follow Up | 22.06 (12.47) | 22.13 (11.87)

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 1 week for each participant.
Description: The definitions are the same as clinicaltrials.gov.
Arm/Group | Imaginal Exposure Writing | Neutral Writing
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/17 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT03734705/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT03734705/ICF_001.pdf